CLINICAL TRIAL: NCT06383988
Title: Multi-Site Community Oncology Planning for the CONNECT Intervention Targeting Lung Cancer Caregivers
Brief Title: A Web-based Program to Help Caregivers of Lung Patients Learn About Available Supportive Care Resources
Acronym: CONNECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00112187; NCI-2023-10870 (Other: NCI Trial Identifier); Lead Organization Identifier (Other: WF-2301CD)
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Stage II Lung Cancer; Stage III Lung Cancer; Stage IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Palliative Care; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Standard care followed by generic resource list) (Active Comparator): Caregivers receive standard care and are then given a generic resource list at week 24.
  Interventions: Other: Support for Caregiver - Generic List
- Group 2 (Generic resource list) (Active Comparator): Caregiver receive a generic resource list at the start of the study.
  Interventions: Other: Support for Caregiver - Generic List
- Group 3 (CONNECT, personalized list, and navigation) (Experimental): Caregivers receive access to the CONNECT tool, watch an educational video on self care and receive a personalized list of resources based on caregiver preferences. Caregivers also receive access to and complete at least 2 calls, at baseline and at week 4, with a caregiver navigator to review the resource list and address any additional needs.
  Interventions: Other: Support for Caregiver - Personalized List; Other: Internet-Based Intervention - CONNECT; Behavioral: Patient Navigation

INTERVENTIONS:
Other: Support for Caregiver - Generic List — Receive a generic resource list
  Arms: Group 1 (Standard care followed by generic resource list); Group 2 (Generic resource list)
Other: Support for Caregiver - Personalized List — Receive personalized resource list
  Arms: Group 3 (CONNECT, personalized list, and navigation)
Other: Internet-Based Intervention - CONNECT — Receive access to CONNECT tool
  Arms: Group 3 (CONNECT, personalized list, and navigation)
Behavioral: Patient Navigation — Complete calls with caregiver navigator
  Other Names: Patient Navigator Program
  Arms: Group 3 (CONNECT, personalized list, and navigation)

SUMMARY:
Clinical trial that tests the feasibility of a web based caregiver support resource, along with caregiver navigation sessions for caregivers of patients with stage II-IV lung cancer. The Caregiver Oncology Needs Evaluation Tool (CONNECT) is a novel web-based intervention designed for the community oncology setting, to systematically connect lung cancer caregivers with tailored supportive care resources. Lung cancer caregivers provide critical and challenging care for their loved ones and are at risk for their own negative psychosocial and physical outcomes. Implementing the CONNECT program along with caregiver navigation may provide additional support to caregivers of patients with stage II-IV lung cancer.

DETAILED DESCRIPTION:
This study is a multi-site randomized pilot trial enrolling 120 lung cancer caregiver-patient dyads (i.e., lung cancer caregivers (n=120) and their care-recipients (n=120)) across approximately 8-12 practices to assess the multi-site feasibility of a caregiver technology-based intervention (CONNECT) to identify caregivers' needs and connect them with supportive care resources. Caregivers will be randomized 1:1:1 to either the CONNECT intervention, usual care comparison group or generic resource list comparison group. CONNECT is a web-based intervention that empowers and educates caregivers about the benefits of supportive care services and systematically identifies unmet needs to connect lung cancer caregivers with tailored supportive care resources. The Central Caregiver Navigator will assist caregivers with resolving barriers to accessing resources and work with the Local Practice Referral Coordinator to process referrals. Caregivers and patients will complete measures at baseline (prior to caregiver randomization), and 12 and 24 weeks after baseline. Feasibility measures (retention, accrual rates, and participation) will be evaluated to inform the future trial. The Local Practice Referral Coordinator for each practice will report on time needed for practice participation, referral processes, and communication processes with the Central Caregiver Navigator.

Participants (i.e., patients or care-recipients) will be asked to complete study surveys at three time points:

* After consenting and before randomization of participant and caregiver. (Initial survey)
* Approximately 12 weeks after completing the first survey (12-week survey)
* Approximately 24 weeks after completing the first survey (24-week survey)

Each survey will take about 30-45 minutes to complete. The forms will ask about things such as demographics (sex, race, etc.), cancer symptoms, satisfaction with cancer care and health behaviors. You don't have to answer any question that makes you feel uncomfortable. These surveys can be done remotely over the internet, in the clinic, by phone or by mail.

Caregivers will also complete surveys at three time points and will be assigned to 1 of 3 study groups:

* Group 1 will be given the usual care provided at your clinic. At the completion of the study, this group will be given the generic supportive care resource list for their use that Group 2 received.
* Group 2 will be provided with a generic supportive care resource list.
* Group 3 will be asked to watch a brief video and complete the web-based CONNECT program either in the clinic or on your own device. The CONNECT program is designed to help identify any unmet needs and connect the caregiver with tailored supportive care resources, based on specific needs. The CONNECT Navigator will follow-up with within 2 business days of completion of the program and again 4 weeks later.

Caregiver Participants (Group 1, 2 and 3) will be asked to complete study surveys at three time points:

* After consenting and before randomization of participant and caregiver. (Initial survey)
* Approximately 12 weeks after completing the first survey (12-week survey)
* Approximately 24 weeks after completing the first survey (24-week survey)

Each survey will take about 35-45 minutes to complete. The forms will ask about things such as demographics (sex, race, etc.), caregiving experience, use of supportive care resources, quality of life, mood, and social needs (housing, transportation, utilities, etc). You don't have to answer any question that makes you feel uncomfortable.

ELIGIBILITY:
Patient Inclusion Criteria:

* Must be ≥ 18 years of age, as this study is focused on the experience of adult patient-caregiver dyads
* Must have a current diagnosis of new (i.e., initial diagnosis) or recurrent stage II-IV lung cancer
* Must be enrolled after the start of anticancer systemic therapy (+/- radiation therapy) with at least 9 weeks of any planned anticancer treatment remaining
* Must be ambulatory and up (i.e., not bedridden) more than 50% of waking hours
* Must self-report receiving informal (i.e., not professional) care from a caregiver who meets the study caregiver criteria and who is willing to participate

Caregiver Inclusion Criteria:

* Must be ≥18 years of age, as this study is focused on the experience of adult patient-caregiver dyads
* Must self-report providing informal (i.e. not professional) care during cancer treatment for a patient who meets the patient criteria and who is willing to participate
* Must have access to the internet at home or be willing to use CONNECT in the clinic
* Must have access to telephone to complete sessions with the central caregiver navigator

Patient Exclusion Criteria:

* Patients who have completed treatment for their lung cancer at the time of study enrollment
* Enrolled in hospice care
* Unable to read and English and not willing to have someone read surveys for them

Caregiver Exclusion Criteria:

* Self-report currently receiving cancer treatment
* Unable to read and communicate in English, as the CONNECT intervention is currently only available in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver retention at 12 weeks | At 12 weeks
  Calculated as the following: Number of caregivers who complete at least 75% of the 12-week assessments divided by the number randomized. Retention will be estimated and reported along with an exact 95% confidence interval.

SECONDARY OUTCOMES:
Caregiver accrual rate | Upon completion of recruitment, approximately 12 months
  Number of caregivers who agree to participate divided by the number of months of recruitment
Caregiver participation | Upon completion of recruitment, approximately 12 months
  Proportion of eligible caregivers who agreed to participate
Caregiver retention at 24 weeks | At 24 weeks
  Number of caregivers who complete at least 75% of the 24-week assessments divided by the number randomized.
Caregiver acceptability | At 12 weeks
  Self-report survey developed for this study to assess the degree to which caregivers found different aspects of CONNECT, the generic resource list, or usual care helpful using a Likert response from 0 (Not at all) to 5 (Very Much)
Average time (minutes) needed for training for Local Practice Referral Coordinator | At completion of training, up to 6 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range.
Desired modality for training (e.g., live webinar, recorded video, paper materials) for Local Practice Referral Coordinator | At completion of training, up to 6 months
  Will be summarized using appropriate descriptive statistics.
Average time (minutes) needed to identify and enter local resources into the Caregiver Oncology Needs Evaluation Tool (CONNECT) database | At conclusion of practice intervention activities, an average of 18 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range.
Frequency of needed resource updates in the CONNECT database | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range
Average time (minutes) spent by the Central Caregiver Navigator and Local Practice Referral Coordinators with each caregiver in the CONNECT arm | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range.
Modality of contact (e.g. phone, virtual web meeting, email) made by the Central Caregiver Navigator and Local Practice Referral Coordinators with each caregiver in the CONNECT arm | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized using appropriate descriptive statistics.
Number of contacts made by the Central Caregiver Navigator and Local Practice Referral Coordinators with each caregiver in the CONNECT arm | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range.
Number of referrals facilitated by the Local Practice Referral Coordinator and Central Caregiver Navigator | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range.
Type of referrals (e.g., in person, online) facilitated by the Local Practice Referral Coordinator and Central Caregiver Navigator | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized using appropriate descriptive statistics.
Average time (minutes) needed to communicate for Central Caregiver Navigator and Local Practice Referral Coordinator | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized across practices using mean, median, standard deviation and interquartile range.
Modalities used for communication (e.g., phone, virtual web meeting, email) for Central Caregiver Navigator and Local Practice Referral Coordinator | Up to completion of practice intervention activities, an average of 18 months
  Will be summarized using appropriate descriptive statistics.
Improvements for the future trial from Local Practice Referral Coordinator's perspectives from a survey at the end of the study | At completion of practice intervention activities, an average of 18 months
  Will be summarized using appropriate descriptive statistics.

OTHER OUTCOMES:
Patient accrual rate | Upon completion of recruitment, approximately 12 months
  Number of patients who agree to participate divided by the number of months of recruitment
Patient participation rate | Upon completion of recruitment, approximately 12 months
  Proportion of eligible patients who agreed to participate
Patient retention at 12 weeks | At 12 weeks
  Number of patients who complete at least 75% of the 12-week assessments divided by the number randomized
Patient retention at 24 weeks | At 24 weeks
  Number of patients who complete at least 75% of the 24-week assessments divided by the number randomized

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, Study Chair — Wake Forest University Health Sciences
Locations (25):
- United States (25):
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Kaiser Permanente - Rock Creek, Lafayette, Colorado
  - Kaiser Permanente - Lone Tree, Lone Tree, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Lake Regional Hospital, Osage Beach, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Wake Forest NCORP Research Base, Winston-Salem, North Carolina
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu
URL: https://nctn-data-archive.nci.nih.gov/